CLINICAL TRIAL: NCT03195270
Title: Use of [18F]FDG PET/MRI in the Diagnosis of Pain Generators and/or Sites of Inflammation and to Monitor Treatment Effects in Patients With Chronic Pain
Brief Title: Use of PET/MR Imaging in Chronic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Feliks Kogan, Assistant Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-24972
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: Positron emission tomography; Magnetic Resonance Imaging; PET/MRI; Fluorodeoxyglucose; FDG; Pain; Chronic Pain; Neuropathic Pain; Inflammatory Pain; Nociceptive Pain
MeSH Terms: conditions — Chronic Pain; Pain; Neuralgia; Nociceptive Pain | interventions — Fluorodeoxyglucose F18; Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants will be recruited based on established criteria for chronic pain. For the PET/MRI scan, the participants will be injected with 10 mCi±1 mCi of [18F]FTC-146 via the antecubital vein in a bolus injection. PET and MRI scans will be acquired simultaneously using a hybrid PET/MRI scanner. Following the scan, participants will be contacted to check for adverse drug events, and any events will be recorded in the case report. The biodistribution of radiotracer will be analyzed using regions of interest (ROI) marked on anatomical structures on magnetic resonance images and quantifying the signal in PET images within the same ROIs. Pharmacokinetic information will be derived using mathematical modeling. Data from chronic pain patients will be compared to historical data from asymptomatic controls.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): [18F]FDG PET/MRI
  Interventions: Drug: [18F]FDG; Device: PET/MRI

INTERVENTIONS:
Drug: [18F]FDG — 10 mCi of [18F]FDG via the antecubital vein in a bolus injection
  Other Names: [18F]Fluorodeoxyglucose
Device: PET/MRI — PET/MRI hybrid scanner used as diagnostic device
  Other Names: Positron emission tomography/magnetic resonance imaging

SUMMARY:
The investigators are studying the ability of PET/MR imaging (using the PET tracer [18F]FDG) to objectively identify and characterize pain generators in patients suffering from chronic pain.

DETAILED DESCRIPTION:
The diagnosis and management of chronic and neuropathic pain syndromes remains a major clinical challenge, and this failure is partly attributed to our inability to identify the hypersensitive and inflammatory changes in the pain-sensing part of our nervous system that is thought to contribute to these syndromes. The lack of a specific, objective diagnostic test for chronic and neuropathic pain syndromes can result in a delay of diagnosis and suboptimal management decisions. This delay in diagnosis is quite unfortunate since the early diagnosis and treatment of a disease is attributed to the highest probability of remission in certain chronic pain syndromes. Additionally, identifying the correct source of pain is of paramount importance since the clinical course and therapeutic interventions are different depending on cause.

Evidence in the literature points strongly toward an active inflammatory component in chronic pain. For example, soft tissue and bony inflammation is known to be an important pathophysiological mechanism for the symptoms of certain neuropathic pain syndromes. Similarly, individuals suffering from chronic sciatica or radiculopathy may suffer from a combination of inflammation and compression of lumbar or cervical spinal nerves. It is also established that inflammatory lesions have increased metabolism and energy requirements and, therefore, are more glucose-avid than normal tissues, showing increased uptake of radiolabeled glucose analogs, such as [18F]fluorodeoxyglucose ([18F]FDG). Correspondingly, [18F]FDG positron emission tomography-magnetic resonance imaging (PET/MRI) represent leading FDA-approved clinical imaging modalities to longitudinally study metabolic changes in the nervous system and non-neural tissues (e.g., muscle, blood vessels, joints, bone, scar tissue, etc.) in patients with chronic pain conditions. One of the goals of the study is to determine whether [18F]FDG PET/MRI can identify sources of inflammation with greater sensitivity, accuracy and objectivity than current diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Chronic pain lasting greater than 2 months. For example: Low back pain, sciatica, complex regional pain syndrome, peripheral nerve injury, fibromyalgia, neuropathy, osteoarthritis, cancer pain, persistent post-operative pain, and migraine.
* Provides informed consent
* On a typical day, pain level of at least 4/10 on a 0-10 Comparative Pain Scale
* Covid Vaccination status: Vaccinated or unvaccinated subjects who received a negative test result from the Covid test within 72 hours of the scan.

Exclusion Criteria:

* MRI-incompatible
* Diabetes
* Pregnant or nursing
* Non-English speaker
* Claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
[18F]FDG PET/MRI as a spatial biomarker for chronic pain | 5 years
  Identification of structures with increased [18F]FDG uptake (SUVmax) corresponding to pain.

SECONDARY OUTCOMES:
[18F]FDG Biodistribution in Healthy Subjects | 5 years
  We will use PET/MRI to establish the normal range of [18F]FDG uptake. (SUVmax) in various anatomic structures, such as the spinal cord, peripheral nerves, dorsal root ganglia, muscle, bones, joints, blood vessels, of asymptomatic subjects.
36 point Study Short-Form Health Survey | 5 years
  Patient-reported state of health.
Oswestry Disability Index | 5 years
  Measure of disability, quality of life.
Visual Analog Scale | 5 years
  A visual, semi-quantitative method for patient-derived self-assessment of pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Feliks Kogan, PhD, Principal Investigator — Assistant Professor of Radiology
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share the individual participant data with other researchers outside our group of researchers or referring physicians.

REFERENCES:
- [Background] Behera D, Jacobs KE, Behera S, Rosenberg J, Biswal S. (18)F-FDG PET/MRI can be used to identify injured peripheral nerves in a model of neuropathic pain. J Nucl Med. 2011 Aug;52(8):1308-12. doi: 10.2967/jnumed.110.084731. Epub 2011 Jul 15. PMID 21764788
- [Background] Do BH, Mari C, Tseng JR, Quon A, Rosenberg J, Biswal S. Pattern of 18F-FDG uptake in the spinal cord in patients with non-central nervous system malignancy. Spine (Phila Pa 1976). 2011 Oct 1;36(21):E1395-401. doi: 10.1097/BRS.0b013e31820a7df8. PMID 21311407
- [Derived] Yoon D, Fast AM, Cipriano P, Shen B, Castillo JB, McCurdy CR, Mari Aparici C, Lum D, Biswal S. Sigma-1 Receptor Changes Observed in Chronic Pelvic Pain Patients: A Pilot PET/MRI Study. Front Pain Res (Lausanne). 2021 Oct 20;2:711748. doi: 10.3389/fpain.2021.711748. eCollection 2021. PMID 35295458
- [Derived] Yoon D, Xu Y, Cipriano PW, Alam IS, Mari Aparici C, Tawfik VL, Curtin CM, Carroll IR, Biswal S. Neurovascular, Muscle, and Skin Changes on [18F]FDG PET/MRI in Complex Regional Pain Syndrome of the Foot: A Prospective Clinical Study. Pain Med. 2022 Feb 1;23(2):339-346. doi: 10.1093/pm/pnab315. PMID 34718774